CLINICAL TRIAL: NCT07289685
Title: Use a Wearable Devices to Observe Complications of Mobilization for Colorectal Cancer After Surgery
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202102412B0; CMRPG3M2171 (Other Grant/Funding Number: Chang Gung Memorial Hospital, Linkou)
Record Dates: First submitted 2025-08-20; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative Colorectal Cancer Patients with Wearable Device Monitoring: Patients diagnosed with colorectal cancer who underwent minimally invasive surgery. Participants wore a wrist-worn device to monitor postoperative physical activity, heart rate, and sleep for up to 7 days or until discharge.

SUMMARY:
This study aims to help patients recover faster after colorectal cancer surgery by using wearable devices to monitor early movement.

Patients will wear a lightweight wristband that tracks heart rate, sleep, and daily steps after surgery. The goal is to find out if early walking can reduce the chances of complications, shorten hospital stays, and lower medical costs.

Participants will start wearing the device after surgery and continue for about 7 days or until they leave the hospital. During this time, they will also fill out a simple daily observation form. Participation is voluntary, and patients can withdraw at any time without affecting their care.

The study hopes to provide new ways to improve recovery and offer better support to patients after colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing minimally invasive colorectal tumor resection.
2. Aged 20 to 85 years.
3. ECOG score 0-2.
4. Clear consciousness and ability to communicate in Mandarin or Taiwanese (or via family translation).
5. Informed consent provided by the patient or family.

Exclusion Criteria:

1. Patients with acute/chronic psychiatric disorders or cognitive impairment.
2. Patients undergoing traditional open or local resection surgeries.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 20 to 85 years diagnosed with colorectal cancer who underwent minimally invasive surgery at a medical center. Patients must be able to communicate in Mandarin or Taiwanese and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay | Through hospital discharge (an average of 7 days after surgery)
  The number of calendar days from the date of colorectal surgery to the date of hospital discharge, recorded from the hospital electronic medical record.

SECONDARY OUTCOMES:
Postoperative Complications (Clavien-Dindo classification) | Postoperative Day 30
  The occurrence and severity of postoperative complications during hospitalization, graded using the Clavien-Dindo classification system based on medical record review.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to the need to protect patient privacy and confidentiality. Additionally, there are no current plans for secondary analysis or collaboration with external researchers.